CLINICAL TRIAL: NCT06627361
Title: Prospective, Multicentric, Comparative, Randomized, Cross-over Study Evaluating the Mobility of Transtibial Amputee Patients Using the PRO-FLEX PIVOT® Foot Versus a Class III Energy Storing and Returning (ESAR) Prosthetic Foot
Brief Title: Comparative Study Evaluating the Mobility of Transtibial Amputee Patients Using the PRO-FLEX PIVOT® Foot Versus a Class III Energy Storing and Returning (ESAR) Prosthetic Foot.
Acronym: DEFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A01374-41
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-01

CONDITIONS: Amputation
Keywords: Lower limb amputation; Mobility; Pro-Flex Pivot; Randomized; ESAR foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRO-FLEX PIVOT (Experimental): The patient will be fitted with PRO-FLEX PIVOT® foot for a duration of 28 days, with a variance of ±2 days
  Interventions: Device: PRO-FLEX PIVOT Foot evaluation
- Class III ESAR foot (Active Comparator): The patient will be fitted with his usual class III ESAR foot for a duration of 28 days, with a variance of ±2 days
  Interventions: Device: Class III ESAR Foot evaluation

INTERVENTIONS:
Device: PRO-FLEX PIVOT Foot evaluation — The subject will wear the PRO-FLEX PIVOT foot for 4 weeks, following which they will complete questionnaires and undergo a Time Up and Go test
  Arms: PRO-FLEX PIVOT
Device: Class III ESAR Foot evaluation — The subject will wear his usual Class III ESAR Foot foot for 4 weeks, following which they will complete questionnaires and undergo a Time Up and Go test
  Arms: Class III ESAR foot

SUMMARY:
The PRO-FLEX PIVOT® is ESAR prosthetic foot with an innovative technology built around three pillars:

1. The PIVOT technology: three axes of rotation (upper support, main pivot and lower support) at the ankle, which allow both a movement with more amplitude and closer to the physiological movement of the ankle, and an increase in the power of the ankle, especially in the terminal support phase.
2. The technology of the three carbon blades (plantar, upper and median), including a wider plantar blade, split in the middle of the foot with a separate toe to provide efficiency over the entire length to the big toe, bringing more power to the impulse and more control, but also increased stability until the terminal support phase.
3. An anatomical foot cosmetic, to adapt and optimize the function of the blade: of light manufacture, with an adherent sole for more stability barefoot, it guarantees physiological plantar pressure during the unwinding of the foot.

The aim of this study is to demonstrate that compared to a class III ESAR foot, the PRO-FLEX PIVOT® foot improves patient mobility with a validated score.

ELIGIBILITY:
Inclusion Criteria:

Adult patient (over 18 years of age)

* Unilateral tibial amputee and fitted for at least 6 months with a class III ESAR foot.
* Regularly using (more than 8 hours/day) a class III ESAR foot
* Functional class (CNEDiMTS indication)1
* Insured person.
* Able to answer questionnaires.
* Providing informed and written consent to participate in the study.
* Having a normalized PLUS-M/FC 12 score less than 50 for vascular amputee and 55 for traumatic amputee and other causes of amputation.
* Experiencing no discomfort related to the socket indicated by a score ≥ 6 on the numerical scale from 0 to 10 (Socket Comfort Score)

Exclusion Criteria:

* Bilateral lower limb amputation
* Femoral amputation
* Wearing a temporary prosthesis
* Change of socket or suspension system planned during the study.
* Change of any functional component as torsion or choc adapter
* Significant change in the patient's routine activities expected during the study.
* Progressive associated pathology that may prevent patient follow-up.
* Associated pathology that may limit the patient's mobility (e.g. disarticulation of the knee, knee pain... )
* No osteointegration patients
* Lack of consent
* Adult subject to enhanced protection, deprived of liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social institution for purposes other than research.
* Person not affiliated with or a beneficiary of a health insurance plan.
* Patient unable to understand the study instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of mobility of the patient | 28 days
  Assess the foot impact on the patient mobility assessed with Prosthetic Limb Users Survey of Mobility (PLUS-M™) questionnaire. The score ranges from 21.8 (indicated lower mobility) to 71.4 (indicating higher mobility)

SECONDARY OUTCOMES:
Variations in comfort experienced during the wearing of the foot | 28 days
  Evaluate the impact of the foot on the comfort experienced by the patient with visual analog scale (VAS) from 0 (= not at all comfortable) to 5 (=Very comfortable)
Change in quality of life | 28 days
  Evaluate the impact of the foot on the quality of life assessed by the Orthotics Prosthetics Users Survey (OPUS) patient Self report questionnaire. The higher the score [0-92], the better the perception of quality of life.
Change in satisfaction of the patient | 28 days
  Assess the change in patient satisfaction with Quebec User Evaluation of Satisfaction with assistive Technology (QUEST = ESAT in French); Higher scores indicate greater satisfaction.
Occurence of falls | 28 days
Number of patients with technical incidents | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Noël MARTINET, PhD, Principal Investigator — IRR - Établissement de Nancy - Louis-Pierquin
Locations (1):
- Multiples locations, Multiple Locations, France

IPD SHARING:
Plan to Share IPD: No